CLINICAL TRIAL: NCT07188402
Title: Sleep Disturbance Prevalence In Bullous Pemphigoid Patients
Brief Title: Prevalence of Sleep Disturbances in Bullous Pemphigoid Patients.
Acronym: SLEEP-BP
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/088/OB; 2020-A00837-32 (Other: ANSM)
Record Dates: First submitted 2025-09-17; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-03

CONDITIONS: Bullous Pemphigoid (BP)
Keywords: Sleep Disturbance Prevalence
MeSH Terms: conditions — Pemphigoid, Bullous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Prevalence of sleep disturbances in patients with bullous pemphigoid — Use of a questionnaire assessing the Insomnia Severity Index (ISI)
Other: Prevalence of sleep disturbances in healthy volunteers without bullous pemphigoid — Use of a questionnaire assessing the Insomnia Severity Index (ISI)

SUMMARY:
Bullous pemphigoid (BP) is the most common autoimmune blistering disorder. The incidence of BP has increased due to increased life expectancy, particularly in developed countries, which can be associated with multiple geriatric comorbidities and polypharmacy.

Epidemiological studies of BP have shown that the incidence ranges from 2.5 to 42.8 cases/million/year in European countries.

BP affects older adults with multiple comorbidities, primarily neurological diseases such as multiple sclerosis, dementia, Parkinson's disease, epilepsy, and stroke, which are usually diagnosed before BP.

Diagnosis is based on clinical suspicion combined with immunopathological investigations. The clinical chronological course is characterized by relapses and remissions. The goals of PB treatment are to stop the development of new skin lesions, healing of old lesions, and symptomatic therapy.

DETAILED DESCRIPTION:
The patient's physical and psychological state can be seriously affected by the disease itself or by the side effects of treatment. These effects could lead to a decrease in the patient's functional capacity and increase the burden, stress, and isolation of the patient and their family. These significant effects may be underestimated by healthcare professionals, which may be partly explained by the paucity of published reports on this particular problem.

Sleep is a fundamental, restorative, physiological, and neurobiological state that consumes approximately one-third of our lives. Sleep is carefully regulated by multiple processes, including homeostatic sleep and the circadian system. Itching and pain can significantly reduce patients' quality of life and sleep.

BP can be a stressful experience and places a significant burden on patients. Patients often have difficulty coping with new changes in daily tasks. Specific daily activities such as housekeeping, dressing, and showering can also be complicated. As a result, patients may experience frustration, depression, low self-esteem, and a reduced quality of life.

Furthermore, pain, itching, and discomfort can negatively impact sleep, mood, and enjoyment of life, further contributing to depression and frustration in these patients.

No studies have been published on the effect of bullous pemphigoid on sleep quality or the prevalence of sleep disturbances in bullous pemphigoid patients, except for a recent study published in January 2019 in the journal Clinical and Experimental Dermatology. This study was conducted in Poland and included a total of 31 participants. The researchers assessed sleep quality using a sleep monitor (Actisleep+) worn in the dominant hand. This study confirmed that PB patients have very poor sleep quality.

Using a patient-centered questionnaire (ISI questionnaire), this study aims to assess the prevalence of sleep disturbances and associated risk factors in patients with bullous pemphigoid. These data will be compared with those of age- and sex-matched control subjects. Control subjects will be recruited from dermatology department consultations and are being monitored for basal cell carcinoma, seborrheic keratosis, actinic keratosis, squamous cell carcinoma, or other benign skin tumors. These dermatological diseases are not known to affect sleep like psoriasis and atopic dermatitis. These control subjects therefore reflect the general population.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Patient
2. Patients: Bullous Pemphigoid: Newly diagnosed by:

   * Rash suggestive of Bullous Pemphigoid
   * Histology: Subepidermal bulla or margination of eosinophils along the dermoepidermal junction (DEJ)
   * Controls: Patient with Basal Cell Carcinoma, Squamous Cell Carcinoma, Seborrheic Keratosis, Actinic Keratosis, or Other Benign Skin Tumor. We selected the control group from these patients because these dermatological conditions do not affect sleep quality.
3. Mini Mental Status Examination (MMS) score > 20
4. No Formulated Opposition

Exclusion Criteria:

1. Protected Adult
2. Advanced Dementia Syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Prospective, non-interventional, descriptive, multicenter case-control study based on a questionnaire (ISI questionnaire) aimed at patients with bullous pemphigoid and healthy volunteers, controls recruited during dermatology department consultations, followed for basal cell carcinoma, seborrheic keratosis, actinic keratosis, squamous cell carcinoma or other benign skin tumor known not to affect sleep.
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
To examine the prevalence of sleep disturbances in patients with bullous pemphigoid compared to a control group using the Insomnia Severity Index (ISI) questionnaire annexed to this protocol. | Enrollment visit and month 1
  The Insomnia Severity Index (ISI), which is a brief instrument designed to assess the severity of both daytime and daytime components of insomnia.
  The total ISI score is interpreted as follows:
  * No insomnia (0-7)
  * Subthreshold insomnia (8-14)
  * Moderate insomnia (15-21)
  * Severe insomnia (22-28)

SECONDARY OUTCOMES:
Determination of disease-related predictors of sleep disorders | Enrollment visit and month 1
  To examine potential disease-related predictors of sleep disorders using the Pemphigus Disease Area Index (BPDAI) score. The Pemphigus Disease Area Index (PDAI) is a standardized clinical tool used to assess the severity and extent of lesions in patients with pemphigus, a rare autoimmune disease that causes bullae (blisters) on the skin and mucous membranes. Score O = Complete remission; Score 1 to 15 mild illness; Score 16 to 45 Moderate disease; score > 46 severe illness.

CONTACTS AND LOCATIONS:
Locations (1):
- University Rouen Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.